CLINICAL TRIAL: NCT05156723
Title: A Double-blind, Randomized, Prospective, Placebo-controlled Trial to Assess the Immunogenicity, Safety, and Tolerability of a Coronavirus Vaccine in Healthy Volunteers Aged 18 to 60 Years
Brief Title: Study of the Immunogenicity, Safety and Tolerability of the Convacell Vaccine.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Collaborators: Crocus Medical B.V (The Netherlands) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01-COVAC-04/21
Record Dates: First submitted 2021-11-26; First posted 2021-12-14 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: COVID-19; Immunologic Factors; Coronavirus Infections; Respiratory Tract Infections
Keywords: COVID-19; COVID; recombinant vaccine; nucleocapsid protein; cellular immunity; SPbSRIVS; Convacell
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1: Subunit recombinant vaccine for the prevention of coronavirus infection (Experimental): 5 volunteers have been vaccinated with a single dose (Stage I)
  Interventions: Biological: Subunit recombinant vaccine for the prevention of coronavirus infection
- Group 2: Subunit recombinant vaccine for the prevention of coronavirus infection (Experimental): 15 volunteers have been vaccinated with a single dose (Stage I)
  Interventions: Biological: Subunit recombinant vaccine for the prevention of coronavirus infection
- Group 3: Subunit recombinant vaccine for the prevention of coronavirus infection (Experimental): 45 volunteers will be vaccinated with the coronavirus vaccine intramuscularly twice (Stage II)
  Interventions: Biological: Subunit recombinant vaccine for the prevention of coronavirus infection
- Group 4: Subunit recombinant vaccine for the prevention of coronavirus infection (Experimental): 45 volunteers have been vaccinated with a single dose of the coronavirus vaccine intramuscularly and then treated with a single dose of placebo (Stage II)
  Interventions: Biological: Subunit recombinant vaccine for the prevention of coronavirus infection
- Group 5: Placebo (Placebo Comparator): 45 volunteers have been vaccinated with placebo intramuscularly twice (Stage II)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Subunit recombinant vaccine for the prevention of coronavirus infection — solution for intramuscular injection, 0.5 ml
  Arms: Group 1: Subunit recombinant vaccine for the prevention of coronavirus infection; Group 2: Subunit recombinant vaccine for the prevention of coronavirus infection; Group 3: Subunit recombinant vaccine for the prevention of coronavirus infection; Group 4: Subunit recombinant vaccine for the prevention of coronavirus infection
Biological: Placebo — solution for intramuscular injection, 0.5 ml
  Arms: Group 5: Placebo

SUMMARY:
A two-stage trial will involve healthy volunteers. The first stage is open trial, and the second stage is a double-blind trial with randomization of volunteers into three groups. At stage I of the trial, the maximum number of screened healthy volunteers will be 30 of which 20 men aged 18 to over 60 years. At stage II of the trial, the maximum number of screened healthy volunteers will be 150, of which 135 men and women aged 18 to over 60 years eligible according to the inclusion and exclusion criteria are planned to be included and randomized to collect data that will be used for the subsequent safety and immunogenicity assessment. The enrollment of volunteers at stage II will be competitive.

DETAILED DESCRIPTION:
Trial product is subunit recombinant vaccine for the prevention of coronavirus infection caused by the SARS-CoV-2 virus.

Vaccination forms humoral and cellular immunity that prevents the development of coronavirus infection caused by the SARS-CoV-2 virus. On the surface of excipients emulsion droplets N-protein is presented to monocytes attracted from the bloodstream due to a local increase in the level of cytokines. Antigen-bearing cells migrate to draining lymph nodes with activation of innate and adaptive immunity cells in them. Due to the activation of natural killer cells in combination with specific antibodies, the mechanism of lysis of infected cells is realized. The nucleocapsid protein (N) is conserved and little susceptible to mutational changes. This makes the vaccine based on it universal for various strains of coronavirus

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women aged 18 to 60 years old, inclusive.
2. Written informed consent of the volunteer to participate in the clinical trial;
3. BMI within the range of 18.5 ≤ BWI ≤ 30 kg/m2 with the body weight of not less than 55 kg for men, not less than 45 kg for women and not more than 100 kg for volunteers of both sexes.
4. Verified "healthy" status: no deviations from reference values of standard clinical, laboratory and instrumental examinations.
5. Negative HIV 1&2, RPR, HВsAg and HCV RNA tests.
6. Hemodynamic and other vital signs are within normal limits (reference intervals are 60-90 beats/min at rest for HR, up to 22 per minute for RR, body temperature from 35.5 to 36.9 °C; systolic blood pressure (SBP) is considered normal in the range of 100-139 mmHg, diastolic blood pressure (DBP) - in the range of 60-89 mmHg);
7. Volunteers able to fulfill requirements of the Protocol (i.e., fill out the patient's diary, come to follow-up visits);
8. Abstinence from alcohol for 14 days before the start of the trial and until the end of participation in the trial;
9. Abstinence from smoking for 48 hours before the start of the trial and during hospitalization;
10. For fertile women - a negative result of the pregnancy test and consent to observe adequate methods of contraception during the trial and at least two months after vaccination;
11. For fertile men - consent to observe adequate methods of contraception during the trial and at least two months after vaccination, except for men after vasectomy with documented azoospermia, and their sexual partners should use methods of contraception that ensure more than 90% reliability or be incapable of conception after a surgical sterilization or have a natural menopause for at least 2 years

Exclusion Criteria:

1. History of influenza or acute respiratory viral infection (ARVI) within 2 months before the start of the trial.
2. A serious post-vaccination reaction (temperature above 40 °C, hyperemia or edema more than 8 cm in diameter) or complications (collapse or shock-like condition that developed within 48 hours after vaccination; convulsions accompanied or not accompanied by a fever due to any previous vaccination).
3. Fever, cough, and shortness of breath within 30 days before vaccination.
4. History of COVID-19.
5. Positive result of the COVID-19 PCR test.
6. Body temperature ≥ 37,0°C.
7. History of allergies.
8. Any vaccination within 30 days before the screening.
9. History of leukemia, tuberculosis, cancer, autoimmune diseases.
10. History of Quincke's edema.
11. Positive blood test results for HIV, syphilis, hepatitis B/C.
12. Volunteers who received immunoglobulin during the last three months before the trial.
13. History of long-term use (more than 14 days) of immunosuppressants or other immunomodulatory drugs for six months before the trial.
14. Treatment with glucocorticosteroids, including in small doses, as well as local use of drugs containing steroids (> 10 mg of prednisolone or its equivalent for more than 14 days before the screening).
15. History of any confirmed or suspected immunosuppressive or immunodeficiency condition.
16. History of splenectomy.
17. History of chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, the gastrointestinal tract, liver, kidneys, hematopoietic or immune systems, mental disease in the acute stage or in the decompensation stage.
18. Transfusion of blood or blood components within 4 months before screening.
19. History of acute and chronic infectious diseases.
20. Consumption of more than 10 units of alcohol per week or history of alcohol addiction, drug addiction or abuse of pharmaceutical products.
21. Smoking of more than 10 cigarettes per day.
22. Participation in another clinical trial within the last 90 days.
23. Pregnancy or lactation.
24. Coagulopathy, hemophilia, bleeding disorder.
25. Participation in stage I of this trial (for volunteers of stage II).
26. Transfusion of COVID-19 convalescent plasma within 14 days before the screening, COVID-19 vaccination less than 30 days before the screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of actively detected local and systemic AEs (Stage I) | During 21 days after initial vaccination
Incidence of actively detected local and systemic AEs (Stage II) | During 21 days after initial vaccination
Increase in geometric mean titers of antibodies to N-protein of SARS-CoV-2 (Stage II) | Days 21 and 42 after the initial vaccination
  Changes from day 0 to days 21 and 42 after the initial vaccination

SECONDARY OUTCOMES:
Incidence of actively detected local AEs | During 7 days after initial vaccination/revaccination
Incidence of actively detected systemic AEs | During 7 days after initial vaccination/revaccination
Incidence of actively detected local AEs | During 21 days after initial vaccination/revaccination
Incidence of actively detected systemic AEs | During 21 days after initial vaccination/revaccination
Incidence of any AEs | During the trial
Number of volunteers hospitalized with COVID-19 | During the trial
  * Total number of SARS-CoV-2 infection cases
  * Total number of COVID-19 cases
  * Total number of COVID-19 related deaths
Proportion SARS-CoV-2 seropositive volunteers | Day 21 (Stage I and Stage II) and Day 42 (Stage II)
Change in IFN-γ, IL-2 and IL-4 levels | Days 14, 21 (Stage I and Stage II) and Days 28, 42, 90 and 180 (Stage II) after vaccination
Change in the subpopulation composition of T-lymphocytes | Days 14, 21 (Stage I and Stage II) and Days 28, 42, 90 and 180 (Stage II) after vaccination
Change in titer of antibodies to N-protein of SARS-CoV-2 | Days 14, 21 (Stage I and Stage II), Days 28, 42, 90 and 180 (Stage II), Days 240, 350 (Stage II, cohort 2) after initial vaccination
Change in the antigen-specific cellular immune response (T-cell response) | Days 14, 21 (Stage II), Days 28, 42, 90 and 180, Days 240, 350 (Stage II, cohort 2) after initial vaccination
Incidence of seroconversion (specific antibodies to N-protein of SARS-CoV-2) | Days 14, 21 (Stage I and Stage II), Days 28, 42, 90 and 180, Days 240, 350 (Stage II, cohort 2) after initial vaccination

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Medvitro, LLC, Moscow
  - Research Institute of Vaccines and Serums them. I.I. Mechnikov, Moscow
  - Eco-Safety, LLC, Saint Petersburg